CLINICAL TRIAL: NCT04228302
Title: A Single-Center, Double-Blind, Placebo-Controlled, Phase 1A Single Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Sequential Dose Regimens of Oral EC5026 in Healthy Male and Female Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Oral EC5026 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EicOsis Human Health Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC5026-1-01; 1UH2NS094258-01 (NIH)
Record Dates: First submitted 2020-01-06; First posted 2020-01-14 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Healthy Adults
MeSH Terms: interventions — EC5026

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EC5026 (Experimental): Single Ascending Doses of oral EC5026
  Interventions: Drug: EC5026 oral capsule
- Placebo (Placebo Comparator): Single doses of matching oral placebo
  Interventions: Other: Placebo oral capsule

INTERVENTIONS:
Drug: EC5026 oral capsule — 5 sequential cohorts of 8 subjects randomly assigned to receive single ascending oral doses of EC5026 (n=6 per cohort) or matching placebo (n=2 per cohort).
  Oral doses of EC5026 tested in each cohort: 0.5 mg (Cohort 1), 2 mg (Cohort 2), 8 mg (Cohort 3), 16 mg (Cohort 4), and 24 mg (Cohort 5).
  A blinded sentinel group of 2 subjects (1 active and 1 placebo) will be dosed at least 2 days before the remaining 6 subjects (5 active and 1 placebo) will receive blinded doses of active study drug or placebo.
  Arms: EC5026
Other: Placebo oral capsule — 5 sequential cohorts of 8 subjects randomly assigned to receive single ascending oral doses of EC5026 (n=6 per cohort) or matching placebo (n=2 per cohort)
  Arms: Placebo

SUMMARY:
This is a first-in-human study with EC5026, a new drug candidate intended to treat neuropathic pain. The purpose of the study is to provide initial safety, tolerability, and pharmacokinetics data of single ascending oral doses of EC5026 in healthy subjects.

DETAILED DESCRIPTION:
This is a single-center, double-blind, placebo-controlled, Phase 1a single ascending dose study evaluating the safety, tolerability and pharmacokinetics of sequential doses of oral EC5026 in healthy male and female subjects. EC5026 is an inhibitor of the soluble Epoxide Hydrolase (sEH) enzyme developed as a first-in-class analgesic for the treatment of pain. This study will help refine the dosing strategy for subsequent multiple-dose studies in healthy subjects and for future clinical trials in patients with neuropathic pain.

sEH is an enzyme that is downstream in the cytochrome P450 (CYP) pathway of the arachidonic acid (AA) cascade. The sEH enzyme is responsible of metabolizing a class of epoxy-fatty acids known as epoxyeicosatrienoic acids (EETs), which are potent, naturally occurring analgesics. EETs are produced at high concentrations in areas of tissue damage and inflammation, but are rapidly metabolized by the sEH enzyme into inactive compounds. Effective inhibition of sEH activity prolongs the ability of EETs to exert their analgesic activity.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. The subject is male of female 18 to 65 years, inclusive
2. The subject is able and willing to provide written informed consent to participate in the study.
3. The subject is considered by the investigator to be in good general health as determined by prestudy medical history, physical examination findings, clinical laboratory test results, and 12-lead electrocardiogram (ECG) results.
4. The subject is willing and able to remain in confinement at the study unit from Day -1 to Day 5 and return to the unit at Days 7 and 14 for additional blood tests and safety evaluations.
5. The subject has a body mass index of 19.0 to 32.0 kg/m2, inclusive, at Screening.
6. The subject has normal blood pressure (systolic blood pressure 90 to 140 mm Hg, diastolic blood pressure 50 to 90 mm Hg), and heart rate (resting heart rate 45 to 90 beats per minute) without medication.
7. The subject has a clinical chemistry profile including electrolytes, alkaline phosphatase (ALP), lactate dehydrogenase, creatine phosphokinase (CPK), creatinine, and urea within the normal range without medication at Screening.
8. The subject has urinalysis results including urinary creatinine within the normal range.
9. The subject is a nonsmoker or is willing to abstain from smoking starting 2 weeks prior to randomization and for the duration of the study.
10. The subject is able to read, understand, and follow the study instructions.
11. Male subjects and their female partners must agree to use double-barrier contraception during the study and for 2 months after receiving the last dose of study drug or provide proof of postmenopausal state (minimum 1 year) or surgical sterility.
12. Male subjects must not donate sperm during the study and for 12 months after receiving the last dose of study drug.
13. Female subjects must be nonpregnant, nonlactating, and either postmenopausal for at least 1 year, or surgically sterile for at least 3 months, or agrees to use double barrier contraception from 28 days prior to randomization and/or their last confirmed menstrual period prior to study randomization (whichever is longer) until 2 months after discharge from the clinic. Female subjects will refrain from using hormonal contraceptives for at least 28 days prior to study entry until the end of study (EOS) visit (Day 14). All female subjects of childbearing potential must have a negative pregnancy test result at Screening and baseline (Day -1).

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. The subject has any abnormalities in any of the following: liver function tests, CPK, or urinalysis results. Liver function tests, CPK, or urinalysis tests may be repeated at the discretion of the investigator, if necessary, to confirm any abnormalities.
2. The subject has used any nonstudy medication(s), including low-dose aspirin for cardiovascular prophylaxis, within 1 week before administration of study drug.
3. The subject has used chemotherapy agents or has a history of cancer, other than nonmetastatic skin cancer that has been completely excised, within 5 years prior to screening.
4. The subject has a history of bacterial, fungal, or viral infection requiring treatment with antibiotics, antifungal agents, or antivirals within 1 month prior to randomization.
5. The subject has a presence or history of peripheral edema within the past 5 years.
6. The subject has a history of congestive heart failure.
7. The subject has used drugs which are CYP inducers or inhibitors within 30 days of randomization (eg, cimetidine, paroxetine, fluoxetine, haloperidol, ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin).
8. The subject has used any dietary aids, supplements, or foods that are known to modulate drug metabolizing enzymes (eg, St. John's wort, grapefruit juice) within 14 days of administration of study drug.
9. The subject has difficulty in swallowing oral medications.
10. The subject has a history of seizure disorder.
11. The subject has serious psychosocial comorbidities as determined by the principal investigator.
12. The subject has cognitive or psychiatric disorders, or any other condition that could interfere with compliance with study procedures and/or confinement in a study unit for 5.5 days.
13. The subject has a history of drug or alcohol abuse within 1 year prior to Screening.
14. The subject has used any other investigational drug within 1 month or 5 half-lives, whichever is longer, prior to randomization.
15. The subject has used prescription drugs within 1 month or 5 half-lives, whichever is longer, prior to randomization.
16. The subject has used over-the-counter medication excluding routine vitamins, but including mega-dose vitamin therapy, within 1 week prior to randomization.
17. The subject has donated and/or received any blood or blood products (more than 450 mL) within 3 months prior to randomization.
18. The subject has a presence or history of active gastrointestinal, renal, hepatic, or coagulant disorder within 1 month prior to randomization.
19. The subject has a presence or history of esophageal or gastroduodenal ulceration within 1 month prior to randomization.
20. The subject has a family history of significant cardiac disease (ie, sudden death in first degree relative; myocardial infarction prior to 50 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EC5026 0.5 mg: Single 0.5 mg dose of oral EC5026
- EC5026 2 mg: Single 2 mg dose of oral EC5026
- EC5026 8 mg: Single 8 mg dose of oral EC5026
- EC5026 16 mg: Single 16 mg dose of oral EC5026
- EC5026 24 mg: Single 24 mg dose of oral EC5026
- Placebo: Single dose of matching oral placebo
Period: Overall Study
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 5 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Continuous [Median (Full Range); unit: years] | 40.5 [30 to 58] | 33.5 [20 to 58] | 28.0 [26 to 62] | 42.0 [25 to 53] | 37.5 [29 to 46] | 45.0 [22 to 57] | 36.0 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 4 | 4 | 5 | 22
  Male | 4 | 3 | 2 | 2 | 2 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 3 | 5 | 4 | 17
  Not Hispanic or Latino | 4 | 5 | 4 | 3 | 1 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 3 | 1 | 0 | 4 | 14
  White | 3 | 3 | 3 | 5 | 6 | 6 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs) [Safety and Tolerability]
Description: All AEs reported or observed during the study will be recorded on the electronic case report forms (eCRF). Information to be collected includes drug treatment, type of event, time of onset, dosage, investigator-specified assessment of severity and relationship to study drug, time of resolution of the event, seriousness, any required treatment or evaluations, and outcome. Any AEs resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. All AEs will be followed until they are resolved, stable, or judged by the investigator to be not clinically significant. The Medical Dictionary for Regulatory Activities will be used to code all AEs. A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in intensity or frequency after exposure.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Any Adverse Events | 2 | 4 | 3 | 6 | 4 | 5
  Any Treatment Emergent Adverse Event (TEAE) | 2 | 4 | 2 | 4 | 4 | 3
  Any Treatment-Related TEAE | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Quantifiable Concentration (AUC 0-t) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the AUC in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026. The PK population will include subjects who received a single dose of EC5026 and have sufficient concentration data to support accurate estimation of at least 1 PK parameter. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: Plasma concentrations following EC5026 0.5 mg were below the limit of quantification for all subjects at all timepoints. For 2 subjects in the EC5026 2 mg dose group, plasma concentrations were quantifiable in fewer than 3 samples. These subjects were excluded from the PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 4 | 6 | 6 | 6 | 0
ng*h/mL |  | 258 (145.4) | 3450 (28.4) | 6780 (23.1) | 9030 (22.1) |

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the Cmax in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026. The PK population will include subjects who received a single dose of EC5026 and have sufficient concentration data to support accurate estimation of at least 1 PK parameter. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: Plasma concentrations following EC5026 0.5 mg were below the limit of quantification for all subjects at all time points. For 2 subjects in the EC5026 2 mg dose group, plasma concentrations were quantifiable in fewer than 3 samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 4 | 6 | 6 | 6 | 0
ng/mL |  | 4.69 (45.8) | 82.7 (11.1) | 220 (16.2) | 301 (14.6) |

4. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the Tmax in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026. The PK population will include subjects who received a single dose of EC5026 and have sufficient concentration data to support accurate estimation of at least 1 PK parameter. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 4 | 6 | 6 | 6 | 0
hours |  | 1.25 [1.25 to 1.30] | 1.25 [1.25 to 1.30] | 1.25 [1.25 to 1.25] | 1.25 [1.25 to 1.25] |

5. Primary Outcome: Terminal Phase Half-life in Plasma (t1/2) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the t1/2 in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026. The PK population will include subjects who received a single dose of EC5026 and have sufficient concentration data to support accurate estimation of at least 1 PK parameter. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: Plasma concentrations following EC5026 0.5 mg were below the limit of quantification for all subjects at all time points. For 2 subjects in the EC5026 2 mg dose group, plasma concentrations were quantifiable in fewer than 3 samples. Given that plasma concentrations for the 2 mg dose group were near the limit of quantification, the estimates for t½ should be viewed with caution.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 4 | 6 | 6 | 6 | 0
hours |  | 143 (63.3) | 59.1 (19.0) | 44.8 (14.0) | 41.8 (14.6) |

6. Primary Outcome: Apparent Total Body Clearance (CL/F) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the CL/F in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026. The PK population will include subjects who received a single dose of EC5026 and have sufficient concentration data to support accurate estimation of at least 1 PK parameter. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: Values for CL/F were excluded from summary statistics when %AUCextrap was >20%. Plasma concentrations following EC5026 0.5 mg were below the limit of quantification for all subjects at all time points. For 2 subjects in the EC5026 2 mg dose group, plasma concentrations were quantifiable in fewer than 3 samples.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 0
L/h |  |  | 2.23 (0.56) | 2.35 (0.52) | 2.62 (0.54) |

7. Primary Outcome: Apparent Volume of Distribution Based on the Terminal Elimination Rate Constant in Plasma (Vz/F) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the Vz/F in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026.
  The PK population will include subjects who received a single dose of EC5026 and have sufficient concentration data to support accurate estimation of at least 1 PK parameter. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: Plasma concentrations following EC5026 0.5 mg were below the limit of quantification for all subjects at all time points. For 2 subjects in the EC5026 2 mg dose group, plasma concentrations were quantifiable in fewer than 3 samples. Values for Vz/F were excluded from summary statistics when %AUCextrap was >20.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 0
liters |  |  | 178 (21.0) | 146 (34.5) | 153 (40.2) |

8. Primary Outcome: Renal Clearance (CLR) in Response to Escalating Dose Regimens of Oral EC5026 [Urine Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine CLR in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026.
  Subjects will be excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: Urine is collected for analysis of EC5026 during the following time intervals: before dosing and 0 to 8 hours, 8 to 16 hours, 16 to 24 hours, 24 to 32 hours, 32 to 40 hours, and 40 to 48 hours after dosing
Population: All urine concentrations were below the limit of quantification for the EC5026 0.5 and 2 mg dose groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 0
L/h |  |  | 0.00679 (64.8) | 0.00473 (76.7) | 0.00794 (58.7) |

9. Primary Outcome: Amount of Drug Excreted Unchanged in Urine Within the Time Interval 0 to 48 (Ae 0-48) in Response to Escalating Dose Regimens of Oral EC5026 [Urine Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the Ae in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026.
  Subjects will be excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: as for outcome 8
Population: All urine concentrations were below the limit of quantification for the EC5026 0.5 and 2 mg dose groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 0
mg |  |  | 0.0127 (65.9) | 0.0210 (86.2) | 0.0487 (70.9) |

10. Primary Outcome: Fraction of Eliminated Dose in Urine From 0 to 48 Hours (Fe 0-48%) in Response to Escalating Dose Regimens of Oral EC5026 [Urine Pharmacokinetics].
Description: Standard noncompartmental methods will be used to determine the Fe% in response to single oral doses of 0.5, 2, 8,16, and 24 mg of EC5026. Subjects were excluded from the PK population when there were fewer than 3 quantifiable plasma samples.
Time Frame: as for outcome 8
Population: All urine concentrations were below the limit of quantification for the EC5026 0.5 and 2 mg groups.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of eliminated dose
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 0
percentage of eliminated dose |  |  | 0.159 (65.9) | 0.132 (86.2) | 0.203 (70.9) |

11. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC 0-inf) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: as for outcome 2
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48, 72, 84, 96, and 108 hours after dosing
Population: Plasma concentrations following EC5026 0.5 mg were below the limit of quantification for all subjects at all timepoints. For 2 subjects in the EC5026 2 mg dose group, plasma concentrations were quantifiable in fewer than 3 samples. These subjects were excluded from the PK population. Values for AUC0 inf were excluded from summary statistics when %AUCextrap was >20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6 | 0
ng*h/mL |  |  | 3690 (26.3) | 6960 (22.1) | 9310 (21.1) |

12. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 48 Hours After Dosing (AUC 0-48) in Response to Escalating Dose Regimens of Oral EC5026 [Plasma Pharmacokinetics].
Description: as for outcome 2
Time Frame: Predose (0 hour), and at 1.25, 2.25, 4.25, 6.25, 8.25, 12.25, 24, 36, 48 after dosing
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
Number analyzed (Participants) | 0 | 4 | 6 | 6 | 6 | 0
ng*h/mL |  | 119 (59.7) | 1870 (7.9) | 4450 (14.7) | 6130 (13.4) |

ADVERSE EVENTS:
Time Frame: 14 days
Description: A TEAE was defined as any event not present before exposure to study drug or any event already present that worsened in intensity or frequency after exposure. A treatment-related TEAE was defined as a TEAE considered related to the study drug.
Arm/Group | EC5026 0.5 mg | EC5026 2 mg | EC5026 8 mg | EC5026 16 mg | EC5026 24 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 2/6 | 4/6 | 2/6 | 4/6 | 4/6 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EC5026 0.5 mg (N=6) | EC5026 2 mg (N=6) | EC5026 8 mg (N=6) | EC5026 16 mg (N=6) | EC5026 24 mg (N=6) | Placebo (N=10)
Medical device site dermatitis (General disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 3 (3) — Dermatitis related to electrocardiogram electrodes placement
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild COVID-19
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Mild headache
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PPD may not publish any articles or make any presentations relating to the Services provided to EicOsis hereunder with respect to a Project or referring to data, information or materials generated as part of the Services without the prior written consent of EicOsis.

DOCUMENTS (2):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT04228302/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT04228302/SAP_001.pdf